CLINICAL TRIAL: NCT06999421
Title: The Impact of Robot-assisted Digital Education on Prenatal Women's Health Literacy: A Randomized Controlled Trial
Brief Title: The Impact of Robot-assisted Digital Education on Prenatal Women's Health Literacy
Acronym: RADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202309040; N202309040 (Registry Identifier: TMU)
Record Dates: First submitted 2025-05-04; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Two-arm parallel group design: one experimental (robot-assisted) and one control (tablet-based video)
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-Assisted Education Group (Experimental): Participants in this group receive a 30-minute robot-assisted digital health education session about gestational diabetes mellitus (GDM). The robot delivers content using animated videos, emotional facial expressions, gesture recognition, and interactive responses via touch and voice input.
  Interventions: Device: Robot with interactive animations, gesture recognition, and touch/voice-based input
- Tablet-Based Education Group (Control) (Experimental): Participants in this group receive the same 30-minute health education content about GDM via a standard tablet. The video is identical to that in the experimental group but lacks interactive features such as gesture recognition or robot expressions.
  Interventions: Device: Standard tablet (video playback only).

INTERVENTIONS:
Device: Robot with interactive animations, gesture recognition, and touch/voice-based input — A humanoid educational robot that provides GDM-related content using animated videos, emotional facial expressions, gesture movements, and voice/touch-based interaction. Designed to increase engagement, reduce anxiety, and improve health literacy among pregnant women.
  Arms: Robot-Assisted Education Group
Device: Standard tablet (video playback only). — A standard touchscreen tablet used to deliver pre-recorded educational videos on GDM. This intervention provides passive viewing without any robot interaction or feedback.
  Arms: Tablet-Based Education Group (Control)

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a robot-assisted digital education program for pregnant women diagnosed with gestational diabetes mellitus (GDM). The intervention aims to reduce anxiety, improve health literacy, and increase satisfaction and acceptance of digital health technologies. Participants are randomly assigned to either a robot-assisted education group or a conventional tablet-based video education group. Outcome measures include anxiety scores, health literacy scores, and educational satisfaction.

DETAILED DESCRIPTION:
This study implemented a robot-assisted digital education method for teaching about gestational diabetes mellitus (GDM) that was intended to reduce anxiety and encourage healthy behaviors among pregnant women. A randomized controlled trial was conducted to assess the effectiveness of the intervention, where 66 pregnant women from a single hospital were randomly assigned to either the experimental group (n = 32) or the control group (n = 34). The experimental group received health education about GDM using a robot, while the control group received the same health education through video presentations on a tablet. The results showed that the implemented robot-assisted digital education method not only reduced anxiety levels among pregnant women, but also influences their health education satisfaction, health literacy, and acceptance of technology. In the global information age, this study can serve as a reference for educators and researchers at medical institutions interested in tracking long-term health education through technological tools.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥21 years
* Diagnosed with gestational diabetes mellitus (GDM)
* Normal first prenatal ultrasound
* Taiwanese nationality
* Provided informed consent

Exclusion Criteria:

* Non-Taiwanese nationality
* Chronic disease history
* Cognitive impairment or psychiatric disorder
* Declined participation

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Anxiety Level | Immediately post-intervention
  Anxiety levels were assessed using a Likert-type scale ranging from 1 (no symptoms) to 5 (severe anxiety).
Health Literacy | Immediately post-intervention
  Health literacy, which also used a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree)

SECONDARY OUTCOMES:
Health education Satisfaction | Immediately post-intervention
  Health education satisfaction was using a Likert scale ranging from 1 (very satisfied) to 5 (very dissatisfied)
Technology Acceptance | Immediately post-intervention
  technology acceptance of the pregnant women was measured using another Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree)

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing Department, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang CL, Xu ZY, Chang CY. The Impact of Robot-Assisted Digital Education on Prenatal Women's Health Literacy: A Randomized Controlled Trial. J Nurs Manag. 2025 Jun 5;2025:8865606. doi: 10.1155/jonm/8865606. eCollection 2025. PMID 40510888
- See also: https://orcid.org/0000-0002-3146-2270 — https://orcid.org/0000-0002-3146-2270

DOCUMENTS (1):
  • Study Protocol (2025-05-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT06999421/Prot_000.pdf